CLINICAL TRIAL: NCT01172314
Title: Effects of Essential Amino Acid Intake on Net Protein Synthesis in Weight-losing Non-small Cell Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 112254
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Weight loss; protein metabolism; essential amino acid intake
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EAA+LEU vs total AA (Experimental)
  Interventions: Dietary Supplement: EAA+LEU vs total AA
- Total AA vs EAA+LEU (Experimental)
  Interventions: Dietary Supplement: Total AA vs EAA+LEU

INTERVENTIONS:
Dietary Supplement: EAA+LEU vs total AA — 15 g as a bolus
  Arms: EAA+LEU vs total AA
Dietary Supplement: Total AA vs EAA+LEU — 15 g as a bolus
  Arms: Total AA vs EAA+LEU

SUMMARY:
Weight loss commonly occurs in lung cancer patients, negatively influencing their quality of life, treatment response and survival. Gains in lean body mass are difficult to achieve in cancer unless specific metabolic abnormalities are targeted. It is our hypothesis that a nutritional supplement containing a high amount of essential amino acids will target the metabolic alterations of cancer patients. Preliminary research performed in our laboratory in elderly supports this hypothesis. We hypothesize that intake of an essential amino acid nutritional supplement will positively influence protein synthesis rate in advanced non-small cell lung cancer (NSCLC) patients. Furthermore, insight in the underlying mechanism of the higher anabolic response of the essential amino acid supplement will be examined. This information will potentially enable us to formulate a supplement that is more effective than normal food intake, and that will reduce the need for muscle protein breakdown.

DETAILED DESCRIPTION:
In this study, we will test the following hypothesis: A high-leucine essential amino acid mixture stimulates whole body protein synthesis (and in this way protein anabolism) to a larger extent than a regular balanced mixture of total (essential and non-essential) amino acids in NSCLC patients with and without recent weight loss. The principal endpoint will be the extent of stimulation of protein synthesis rate as this is the principal mechanism by which either amino acid or protein intake causes muscle anabolism. This project will provide important clinical information, based on novel fundamental basic knowledge on the process and the specific underlying mechanisms of muscle wasting in patients with NSCLC, and the role of EAA as a potential anabolic substrate. In this way, it will provide preliminary data for the development of nutritional strategies that will prevent or even stop this process of ongoing muscle loss in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Recently diagnosed with Stage III (unresectable) or Stage IV lung cancer (only for the NSCLC group)
2. Ability to sign informed consent
3. Age 40 years and older

Exclusion Criteria:

1. Previous anti-cancer therapy (e.g. radiotherapy, chemotherapy) or surgery less than 4 weeks prior to the experiment.
2. Presence of fever within the last 3 days
3. Established diagnosis of Diabetes Mellitus
4. BMI > 35 kg/m2
5. Untreated metabolic diseases including hepatic or renal disorder
6. Presence of acute illness or metabolically unstable chronic illness
7. Use of long-term oral corticosteroids or short course of oral corticosteroids in the preceding month before enrollment
8. Diagnosis of moderate to severe chronic airflow limitation, defined as measured forced expiratory volume in one second (FEV1) ≤ 70% of referen¬ce FEV1 (only for the healthy control group)
9. Use of supplements enriched with amino acids
10. Any other condition according to the PI or study physicians would interfere with proper conduct of the study / safety of the patient
11. Failure to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-07-13 (Actual); Primary Completion 2012-02-22 (Actual); Study Completion 2012-02-22 (Actual)

PRIMARY OUTCOMES:
Acute change in Net whole body protein synthesis rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement

SECONDARY OUTCOMES:
Acute change in Whole body myofibrillar protein breakdown rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in Whole body collagen breakdown rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in Urea turnover rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in Arginine turnover rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in Liver protein synthesis rate | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in plasma Insulin concentrations | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in plasma Amino acid concentrations | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement
Acute change in plasma Glucose concentrations | Up to 2 years
  Acute change from postabsorptive state after intake of essential amino acid + LEU vs total amino acid supplement

CONTACTS AND LOCATIONS:
Overall Officials: Marielle PK Engelen, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Jonker R, Deutz NE, Erbland ML, Anderson PJ, Engelen MP. Alterations in whole-body arginine metabolism in chronic obstructive pulmonary disease. Am J Clin Nutr. 2016 Jun;103(6):1458-64. doi: 10.3945/ajcn.115.125187. Epub 2016 May 4. PMID 27146652
- [Derived] Engelen MPKJ, Safar AM, Bartter T, Koeman F, Deutz NEP. High anabolic potential of essential amino acid mixtures in advanced nonsmall cell lung cancer. Ann Oncol. 2015 Sep;26(9):1960-1966. doi: 10.1093/annonc/mdv271. Epub 2015 Jun 25. PMID 26113648